CLINICAL TRIAL: NCT01709539
Title: Clinical Evaluation of a New Cancer Diagnosis Center at Kristianstad General Hospital, Sweden
Acronym: CPF-DC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CPF-DC
Record Dates: First submitted 2012-10-12; First posted 2012-10-18 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Cancer
Keywords: Cancer diagnosis center; Time to diagnosis; Survival; Health economics; Biomarkers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diagnostiskt Centrum (Experimental): Investigation at the primary care center followed by further investigation at Diagnostiskt Centrum, Kristianstad General Hospital
  Interventions: Procedure: Diagnostiskt Centrum
- Existing diagnostic procedures (No Intervention): Investigation at the primary care center followed by further investigation at Helsingborg General Hospital

INTERVENTIONS:
Procedure: Diagnostiskt Centrum — Patients who are suspected of having cancer after investigation at the primary care center will be referred to Diagnostiskt Centrum. Each patient who is referred to Diagnostiskt Centrum will undergo the following: (1) clinical chemistry/microbiology tests; (2) medical history; (3) objective clinical examination; and (4) taking of blood samples for analysis of biomarkers. If necessary, patients will also undergo the following: (5) additional laboratory tests; (6) biopsy; (7) X-ray of painful joints; (8) CT scan of the neck, thorax, abdomen, and/or pelvis; (9) mammography and gynecological examination; (10); gastroscopy and/or colonoscopy; and (11) further investigation (e.g., PET-CT scan).
  Other Names: Cancer diagnosis center, Kristianstad General Hospital
  Arms: Diagnostiskt Centrum

SUMMARY:
The aim of this study is to evaluate a new cancer diagnosis center (Diagnostiskt Centrum, DC) in Kristianstad, Sweden. Patients aged ≥ 18 years who are suspected of having serious illness but who have no organ-specific symptoms will be referred to the DC for further investigation after preliminary assessment in primary care. The overall purpose of the study is to evaluate whether the DC meets its target time for diagnosing cancer. In addition, we will evaluate secondary issues, such as survival, to determine whether this pilot project merits extension to other parts of southern Sweden.

DETAILED DESCRIPTION:
Diagnostiskt Centrum (DC), Sweden's first specialized cancer diagnosis center, was established at Kristianstad General Hospital in 2012 as a model for reducing the time taken to diagnose cancer in primary care patients with diffuse, non-organ specific symptoms. If it is successful, the DC model could be rolled out to other areas of Sweden. This study by the Center for Primary Health Care Research in Malmö, Sweden and Regionalt cancercentrum syd will investigate whether the DC process reduces the time from (1) the point when the patient first contacts his/her primary care center with symptoms to (2) the point when he/she is informed about his/her diagnosis (of cancer or another disease). This will be achieved by comparison with matched control patients with suspected cancer who will be referred to Helsingborg General Hospital for further investigation according to existing diagnostic procedures. Various outcome measures will be investigated, and patients' experiences of the DC process will be assessed using a tailored questionnaire. In addition, the DC model will be subjected to health economics analysis.

ELIGIBILITY:
Individuals in two cities in southern Sweden (Helsingborg and Kristianstad) who contact their primary care center because of diffuse, non-organ-specific symptoms

Inclusion criteria: suspicion of cancer following preliminary investigation in primary care

Exclusion criteria: (1) age < 18 years; and (2) inability to fill in the patient questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2012-10; Primary Completion 2019-06 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Time from first contact with primary care to information on diagnosis | After completion of investigation at Diagnostiskt Centrum/Helsingborg General Hospital (anticipated to be up to 37 days)
  The time from the point at which the patient first makes contact with his/her primary care center to the point when he/she is given his/her diagnosis. This comprises two elements: (1) investigation in primary care and (2) investigation at Diagnostiskt Centrum/Helsingborg General Hospital. These two elements will be investigated as secondary outcome measures.

SECONDARY OUTCOMES:
Time from first contact with primary care to decision to refer to Diagnostiskt Centrum/Helsingborg General Hospital | After completion of investigation at Diagnostiskt Centrum/Helsingborg General Hospital (anticipated to be 10-15 days)
Time from decision to refer to Diagnostiskt Centrum/Helsingborg General Hospital to information on diagnosis | After completion of investigation at Diagnostiskt Centrum/Helsingborg General Hospital (anticipated to be up to 22 days)
Survival after diagnosis of cancer or another serious disease | For up to 10 years after diagnosis
Sick leave | During the diagnosis process and for 24 months after diagnosis
Health care utilization | During the diagnosis process and for 24 months after diagnosis
Overall medication use | During the diagnosis process and for 24 months after diagnosis
Use of analgesics, antidepressants, and other psychotropic drugs | During the diagnosis process and for 24 months after diagnosis
Time from information on diagnosis to decision about treatment | From information on diagnosis to decision about treatment (anticipated to be up to 2 months)
Time from information on diagnosis to initiation of treatment | From information on diagnosis to decision about treatment (anticipated to be up to 3 months)

OTHER OUTCOMES:
Serum inflammatory biomarker levels | During the diagnosis process (anticipated to be up to 37 days after first contact with primary care)
  Serum inflammatory cytokine levels will be compared between patients diagnosed with cancer and patients not diagnosed with cancer (Diagnostiskt Centrum patients only).
Serum epidermal growth factor (EGF) receptor levels | During the diagnosis process (anticipated to be up to 37 days after first contact with primary care)
  Serum EGF receptor levels will be compared between patients diagnosed with cancer and patients not diagnosed with cancer (Diagnostiskt Centrum patients only).
Plasma microRNA levels | During the diagnosis process (anticipated to be up to 37 days after first contact with primary care)
  Plasma microRNA levels will be compared between patients diagnosed with cancer and patients not diagnosed with cancer (Diagnostiskt Centrum patients only).
Telomere length | During the diagnosis process (anticipated to be up to 37 days after first contact with primary care)
  Telomere length (measured using whole-blood samples) will be compared between patients diagnosed with cancer and patients not diagnosed with cancer (Diagnostiskt Centrum patients only).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sundquist, MD, PhD, Principal Investigator — Center for Primary Health Care Research, Malmö, Sweden
Locations (2):
- Sweden (2):
  - Helsingborg General Hospital, Helsingborg, Skåne County
  - Diagnostiskt Centrum, Kristianstad General Hospital, Kristianstad, Skåne County

REFERENCES:
- [Derived] Sundquist J, Palmer K, Ryden S, Savblom C, Ji J, Stenman E. Time Intervals Under the Lens at Sweden's First Diagnostic Center for Primary Care Patients With Nonspecific Symptoms of Cancer. A Comparison With Matched Control Patients. Front Oncol. 2020 Nov 30;10:561379. doi: 10.3389/fonc.2020.561379. eCollection 2020. PMID 33330029